CLINICAL TRIAL: NCT02498730
Title: Can the High Intensity Interval Training (HIIT) Deliver Superior and Rapid Decrease of Symptoms of Bipolar Disorder? a Controlled and Randomized Study
Brief Title: Interval Training in Bipolar Disorder
Acronym: HIIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Alberto Souza de Sá Filho, Doctorade in Mental Health, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFRJ-01
Record Dates: First submitted 2015-07-11; First posted 2015-07-15 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; VO2max; aerobic exercise
MeSH Terms: conditions — Bipolar Disorder | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Interval Training (Active Comparator): 6 stimulous (30 s) at 100% VO2Max/ 1 min 30 s to rest, 19 minutes (total exercise), 3 times/ week, 12 weeks
  Interventions: Behavioral: Interval Training; Behavioral: Continuous Training
- Continuous Training (Active Comparator): Running at 60% VO2Max, 25 minutes (total exercise), 3 times/week, 12 weeks
  Interventions: Behavioral: Interval Training; Behavioral: Continuous Training
- Control (Sham Comparator): Only Dependent Variables Measures
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Interval Training — High Intensity Interval Training at 100% VO2Max
  Other Names: High intensity interval training; HIIT; HIT
  Arms: Continuous Training; Interval Training
Behavioral: Continuous Training — Continuous Stimulous at 60% VO2Max
  Other Names: Moderate Training; Endurance
  Arms: Continuous Training; Interval Training
Behavioral: Control — Only Dependent Variables Measures
  Other Names: No Intervention
  Arms: Control

SUMMARY:
Our main objective will be to evaluate the chronic effects (12 weeks) of high-intensity interval training compared to moderate intensity (same total work) on reducing the symptoms of bipolar disorder, cortical changes, as well as on the VO2max. In addition, the investigators will establish what influence of gain to VO2max has on reducing symptoms.

DETAILED DESCRIPTION:
Physical exercise has significant effects on health promotion and the consequent reduction of the severity of bipolar disorder (BD). This review establishes a pattern of response of exercise and potential impact on the pathophysiology of BD; , as well as, produces hypotheses on how acute and chronic effect of exercises may act differently; and provides future perspectives with the focus of the exercise as an important and innovative model of treatment for BD and mental disorder. A critical evaluation of the literature was undertaken including the influence of exercise on health promotion in patients with mental disorders, neurochemical behavior exercise-induced, as well as reflective introduction of news perspectives of training control in severe exercise domain. The exercise induces significant changes in monoaminergic after, and with long-term training, and work with a threshold of exercise can modulate positive effects on mood. Fast adaptive effects from the high intensity interval training should be considered in BD patients. However, there must be caution in his administration. We speculate that exercise may be a way of maintaining euthymia in the case of BD, making it less vulnerable patient to stay longer at a time of neutrality. Future research is needed to adopt a training strategy that is both time efficient in the different areas and adequate for the population in question.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar Criteria (DSM-IV),
* sedentary lifestyle

Exclusion Criteria:

* 60 and over,
* Cardiovascular Disease,
* Panic disorder,
* Metabolic syndrome Diagnosis

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-08; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Symptom Scales (Hamilton and Young) | 0 week, 6 week, 12 week
  Variable Measured to reduction of symptoms

SECONDARY OUTCOMES:
Cortical Changes (EEG) - Loreta | 0 week, 6 week, 12 week
  Measured to evaluate changes due to training
VO2Max | 0 week, 6 week, 12 week
  Variable Measured to assess cardiovascular improvement
Cognitive Function | 0 week, 6 week, 12 week
  Executive Function, Time Reaction, Atention, and Memory

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio E. Machado, PhD, Study Director — Universidade Federal do Rio de Janeiro
Locations (1):
- Institute of Psychiatry (IPUB), Rio de Janeiro, Brazil